Cost Effectiveness, Safety, and Efficacy of the Kaneka iED Coil System for the Treatment of Wide Necked Ruptured and Unruptured Intracranial Aneurysms

PI: Tomoyoshi Shigematsu

NCT05636124

Document Date: 3/14/2025

## 

Study ID: STUDY-22-01480 Form Version Date: 5March2025

#### STUDY INFORMATION:

**Study Title:** Cost Effectiveness, Safety, and Efficacy of the Kaneka iED Coil System for the Treatment of Wide Necked Ruptured and Unruptured Intracranial Aneurysms (CLASS)

Study site(s): Icahn School of Medicine at Mount Sinai, Mount Sinai Hospital, Mount Sinai West

Lead Researcher (Principal Investigator): Tomoyoshi Shigematsu, MD, PhD

Physical Address: The Mount Sinai Hospital, 1 Gustave L. Levy Place, New York, NY 10029

Mailing Address: 1468 Madison Avenue, Annenberg Building, 20th Floor – Room 225, New York, NY

10029

**Phone:** 212-241-1547

#### SUMMARY OF THIS RESEARCH STUDY:

This document explains a research study you might be interested in joining. Participation in the study is voluntary. You can agree to join or not. Your decision will not limit your ability to receive care at Mount Sinai. You should only agree to take part if you understand the study and if all of your questions about the research study are answered. If you do join the study, the research team must share any new information with you that may change your mind about taking part.

The purpose of this research study is to investigate the cost and secondary endpoints, effectiveness, safety and performance of the Kaneka i-ED TM coil system in the treatment of both ruptured and unruptured wide neck intracranial aneurysms. The cost of endovascular coils is a major contributor to procedural cost in the treatment of intracranial aneurysms. One potential method for controlling cost is to decrease the number of coils used per case without significantly increasing the cost per coil. The Kaneka iED is a diameter coil that may have the ability to achieve comparable embolization to standard devices while using fewer coils, thus controlling cost.

If you choose to take part, you will be asked to provide informed consent, provide your past medical history, undergo treatment of the target aneurysm with the study device, and follow up 1-7 days, 30 days, 6 months, and 18 months post-operation, while submitting to neurological exams, DSA examinations, and providing information for modified Rankin Scale (mRS) and National Institute of Health Stroke Scale (NIHSS) assessments. When using the Kaneka iED, the standard of care for endovascular intracranial aneurysm embolization will be followed and no additional risks are

-----FOR IRB USE ONLY------

Rev 11.11.2022 (Amendment 1-03.09.2023)



## 


anticipated. You will not be paid for taking part in this study. Being in this study will not cost you anything extra. Researchers will not pay you for your travel or the time it will take for you to be in the study.

If you choose to take part, the main risk to you is the risk of loss of private information; this risk always exists, but there are procedures in place to minimize the risk.

You will not benefit directly from taking part in this research.

Instead of taking part in this research, you may use the Kaneka i-ED coil device to treat your aneurysm, regardless of your participation in this study. There might have been alternate procedures for your medical condition, however, your doctor decided to use the Kaneka iED coil device as the best option for you.

If you are interested in learning more about this study, please continue to read below.

#### STUDY PARTICIPATION:

You may qualify to take part in this research study because you have received a diagnosis of ruptured or unruptured wide-neck intracranial aneurysms, as confirmed by radiographic imaging.

Your participation in this research study is expected to last 18 months (end of the follow-up period).

There are 30 people expected to take part in this research study at the Icahn School of Medicine at Mount Sinai, Mount Sinai Hospital, and Mount Sinai West, and 50 people to take part across all sites.

Funds for conducting this research study are provided by Kaneka, the manufacturer of the study device.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

#### **DESCRIPTION OF WHAT IS INVOLVED:**

If you agree to take part in this research study, here is what may be involved:

Rev 11.11.2022 (Amendment 1-03.09.2023)



### ****


- MRA and/or CTA evaluation
- Provide informed consent
- Review of medical history and medication requirements
- Modified Rankin Scale (mRS) and National Institutes of Health Stroke Scale (NIHSS) assessments
- Treatment of target aneurysm with study device
- Neurological exam

**Future Contact:** 

- o DSA (digital subtraction angiogram) examination
- o Study activities will be conducted within the Mount Sinai Health System
- MRA and/or CTA evaluation

You will have follow-up assessments performed by a qualified member of the research team at Day 1, Day 30 follow up, 6-month follow up, and 18-month follow up appointments. All assessments done at these time points are as per standard of care treatment.

Because this research study involves the use of an investigational medical device, a note must be included in your electronic medical record that you are taking part in the research. This way, anyone involved in your medical care will know that you are a study participant, and they can work to avoid any problems or negative outcomes that could arise if they do not know.

# The researchers may wish to use your personal contact information to contact you in the future. Do you give the researchers permission to contact you in the future to request the collection of additional information about you, discuss how your private information, study data and/or samples might be used, or discuss possible participation in another research study?

| Please initial your o | hoice: Yes | No | | |
|---|---|---|---|---|
| If "Yes", please indi | cate your preferr | ed method of co | ontact: (initial all tha | at apply) |
| [ ] Email | [ ] Phone | [ ] Letter | [] Text | |

#### **USE OF YOUR DATA AND/OR SAMPLES:**

The research team will never use or share your personal information (such as, name, address, date of birth, social security number), study data and/or samples (blood, tissue, urine, saliva, or any other 

Rev 11.11.2022 (Amendment 1-03.09.2023)



### ****


body matter) that are collected as part of this study for future research, even if your identity is removed. Your data and/or samples will only be used to complete this study and then they will be destroyed.

#### YOUR RESPONSIBILITIES IF YOU TAKE PART IN THIS RESEARCH:

If you decide to take part in this research study, you will be responsible for the following things: following your doctor's orders and returning for your scheduled follow-up visits.

#### COSTS OR PAYMENTS THAT MAY RESULT FROM PARTICIPATION:

You will not be paid for taking part in this study. Being in this study will not cost you anything extra. Researchers will not pay you for your travel or the time it will take for you to be in the study.

#### **POSSIBLE BENEFITS:**

This study is not designed to benefit you personally. However, possible future benefits to others include embolization of the target aneurysm with equivalent safety and efficacy to the reference devices, and with the potential for decreased cost.

#### POSSIBLE RISKS AND DISCOMFORTS:

- Risk of loss of private information; this risk always exists, but there are procedures in place to minimize the risk.
- In addition to this risk, this research study may hurt you in ways that are not known. The unknown risks could be minor or major (death).

There are no physical, psychological, social, legal, economic risks as a result of taking part in the study. The technique proposed is equivalent to other techniques.

#### OTHER OPTIONS TO CONSIDER:

You may decide not to take part in this research study. If you decide not to take part, this will not affect the clinical care you receive at Mount Sinai. The choice is totally up to you.

Instead of being in this research study, your choices may include:

-----FOR IRB USE ONLY-----

Rev 11.11.2022 (Amendment 1-03.09.2023)



## 


 Using the Kaneka i-ED coil device to treat your aneurysm regardless of your participation in this study. There might have been alternate procedures for your medical condition, however, your doctor decided to use the Kaneka iED coil device as the best option for you.

#### IN CASE OF INJURY DURING THIS RESEARCH STUDY

If you are injured or made sick from taking part in this study, you will get medical care. The group funding this research study will pay you for any reasonable and necessary medical expenses to diagnose and treat research-related injury or illness. This does not prevent you from seeking payment for injury related to malpractice or negligence. You can contact the Lead Researcher for more information.

The Centers for Medicare and Medicaid Services (CMS) is the government agency that oversees Medicare and Medicaid. Funding agencies who make payments for injuries related to studies must report payments to CMS. In order to do this, the funder must have certain information about you, such as your name, date of birth, Social Security Number, Medicare or Medicaid ID numbers, date of injury, and description of injury. The funding agency is only allowed to use this information to report payments related to the injury should this be necessary or as otherwise specified in the Authorization to Use and Disclose Protected Health Information section, which is included below.

#### **ENDING PARTICIPATION IN THE RESEARCH STUDY:**

You may stop taking part in this study at any time. No matter what you choose, your care and benefits through Mount Sinai will not be negatively impacted.

If you decide to stop being in the study, please contact the Lead Researcher or the research staff.

You may also withdraw your permission for the researchers to use and share any of your protected information for research, but <u>you must do so in writing</u> to the Lead Researcher at the address on the first page. Even if you withdraw your permission, the Lead Researcher may still use the information that was already collected if that information is necessary to complete the research study. Your health information may still be used or shared after you withdraw your authorization if you have an adverse event (a bad effect) from taking part in the research study.

If you decide you don't want your data and/or samples to be used for research anymore, you can contact the researcher and ask to have your data and/or samples withdrawn or labeled so that they will not to be used in additional projects or shared. If your data and/or samples have already been shared with researchers, those researchers will be asked to stop using them. However, if any data

-----FOR IRB USE ONLY------

Rev 11.11.2022 (Amendment 1-03.09.2023)



### 


and/or samples have already been shared without your identity or a linking code, it won't be possible to retrieve them. Data and/or samples that have already been used will not be affected by your decision. If your data and/or samples have already been deposited in an external repository, the study team will request that your data and/or samples be removed.

<u>Withdrawal without your consent</u>: The Lead Researcher, the funder or Mount Sinai may stop your involvement in this research study at any time without your consent. This may be because the research study is being stopped, the instructions of the research team have not been followed, the Lead Researcher believes it is in your best interest, or for any other reason. If data and/or samples have been stored as part of the research study, they too can be destroyed without your consent.

#### **CONTACT INFORMATION:**

If you have any questions, concerns or complaints at any time about this research, or you think the research has harmed you, please contact the office of the research team and/or the Lead Researcher at phone number 212-241-1547.

If there is an emergency, please call 911 or go to the emergency room. Let the emergency room staff know you are in a research study so they can contact the Lead Researcher if needed.

#### **DISCLOSURE OF FINANCIAL INTERESTS:**

Researchers sometimes get paid for consulting or doing work for companies that produce drugs, biologics or medical devices. If you have questions regarding industry relationships, you are encouraged to talk to the Lead Researcher or visit our website at http://icahn.mssm.edu/ where Mount Sinai publicly discloses the industry relationships of our faculty.

The company sponsoring this research study makes the device being tested and has a financial interest that could be affected by the outcome of this research study.

Dr. Tomoyoshi Shigematsu (the Mount Sinai Principal Investigator) is a paid consultant for Kaneka Medical, the study sponsor and manufacturer of the Kaneka iED study device.

Mount Sinai receives compensation from the study sponsor, Kaneka, for Dr. DeLeacy's role as the national Principal Investigator (the physician lead) of this study. Dr. DeLeacy does not receive personal compensation from Kaneka for this role. Dr. DeLeacy also serves as a local co-Investigator at Mount Sinai.

------FOR IRB USE ONLY------

Rev 11.11.2022 (Amendment 1-03.09.2023)



## 


Dr. Shigematsu, Dr. Reade DeLeacy, Dr. Johanna Fifi, Dr. J Mocco, and Dr. Shahram Majidi (co-Investigators in this study) are paid consultants and/or have ownership interests with companies that manufacture devices for the treatment of neurovascular disorders including aneurysms and strokes.

In addition, Dr. Mocco is a manager for Neurotechnology Investors (a company which invests in startup companies).

Dr. Christopher Kellner (a co-Investigator in this study) is founder and equity owner of Metis Innovative, a company that invests in medical devices and technology in the neuroscience field.

If you have questions regarding paid relationships that your physician/researcher may have with industry, we encourage you to talk with him or her, or check for industry relationships posted on individual faculty pages on our website at http://icahn.mssm.edu/.

Researchers and/or their departments receive money from the company sponsoring this research based on how many participants they enroll.

#### **MAINTAINING CONFIDENTIALITY – HIPAA AUTHORIZATION:**

As part of this study, some of your private and/or protected health information will be obtained, used, and shared with your permission. There is a Federal Health Insurance Portability and Accountability Act (HIPAA) that makes sure this is done correctly and safely.

#### What is protected health information (PHI)?

PHI is the combination of two things:

- 1. PHI contains information that identifies you. It will be used to contact you and link you to your health information, like name, date of birth, medical record number, and address.
- 2. PHI also contains health information, including information about your mental and physical health from your visits to doctors or hospitals, or from study visits.

Every time you visit a hospital or your doctor, PHI is created and recorded in your medical record by your healthcare providers. In the same way, the PHI created as part of this study will be linked to who you are and your medical information.

What PHI is collected and used in this research study, and might also be shared with others?

As part of this study, the research team at the hospital(s) involved in the research will collect your name, address, telephone/fax numbers, dates directly related to the individual (birth, admission, discharge, date of death, etc.), e-mail/internet protocol (IP) addresses or web universal resource locators (URL's), social security number, medical records number, health plan numbers.

------FOR IRB USE ONLY------

Rev 11.11.2022 (Amendment 1-03.09.2023)



## 


During the study, the researchers will gather information by:

- Reviewing and/or taking your medical history (includes current and past medications or therapies, illnesses, conditions or symptoms, family medical history, allergies, etc.)
- Doing a physical examination that generally also includes blood pressure reading, heart rate, breathing rate, and temperature.
- Completing the tests, procedures, questionnaires and interviews explained in the description section of this consent.

#### Why is your PHI being used?

Researchers need the information that identifies you so they can contact you during the study. They need your health information and the results of any tests and procedures being collected as part of this study to answer the questions posed in the study. The purpose of the study is discussed earlier in this consent form. Before researchers analyze the data, they remove any information that would let others know who you are or that you took part in the study. If researchers publish or present study results at scientific meetings, lectures, or other events, their presentations would not include any information that would let others know who you are, unless you give separate permission to do so.

The Lead Researcher may also use and share the results of these tests and procedures with other healthcare providers at Mount Sinai who are involved in your care or treatment. The research team and other authorized members of The Mount Sinai Health System ("Mount Sinai") workforce may use and share your information to ensure that the research meets legal, institutional or accreditation requirements. For example:

- The Mount Sinai Program for the Protection of Human Subjects is responsible for overseeing research on human participants and may need to see your information.
- If you receive any payments for taking part in this study, the Mount Sinai Finance Department may need your name, address, social security number, payment amount, and related information for tax reporting purposes.
- If the research team uncovers abuse, neglect, or reportable diseases, this information may be disclosed to appropriate authorities.

#### Who, outside Mount Sinai, might receive your PHI?

As part of the study, the Lead Researcher, research team and others in the Mount Sinai workforce may disclose your PHI, including the results of the research study tests and procedures, to the following people or organizations: (It is possible that there may be changes to the list during this research study; you may request an up-to-date list at any time by contacting the Lead Researcher.)

- The United States Department of Health and Human Services (DHHS) and the Office of Human Research Protection (OHRP) (the government organization that is responsible for protecting human research participants).

------FOR IRB USE ONLY------

Rev 11.11.2022 (Amendment 1-03.09.2023)



## 


- The commercial sponsor and/or their representative (who will use the results for submissions to the Food and Drug Administration (the government organization that approves drugs or devices for medical use): Kaneka.
- Academic Research Organization (whose job is to help organizations fulfill their responsibilities in the research and development process): Mount Sinai Health System.
- A Data Safety Monitoring Board or other committee that will monitor the study on an ongoing basis for safety.
- The United States Food and Drug Administration.

In all disclosures outside of Mount Sinai, you will not be identified by name, social security number, address, telephone number, or any other direct personal identifier unless disclosure of the direct identifier is required by law. Some records and information disclosed may be identified with a unique code number. The Lead Researcher will ensure that the key to the code will be kept in a locked file, or will be securely stored electronically. The code will not be used to link the information back to you without your permission, unless the law requires it, or rarely if the Institutional Review Board (IRB) allows it after determining that there would be minimal risk to your privacy. It is possible that a sponsor or their representatives, a data coordinating office, a contract research organization, may come to inspect your records. Even if those records are identifiable when inspected, the information leaving the institution will be stripped of direct identifiers. Additionally, when applicable, the monitors, auditors, the IRB, OHRP, as well as the Food and Drug Administration (FDA) will be granted direct access to your medical records for verification of the research procedures and data. OHRP and FDA are authorized to remove information with identifiers if necessary to complete their task. By signing this document you are authorizing this access. The results of this research may be published. However, your name and other identifying information will be kept confidential.

<u>For how long will Mount Sinai be able to use or disclose your PHI?</u> Your authorization for use of your PHI for this specific study does not expire.

#### Will you be able to access your records?

During your participation in this study, you will have access to your medical record and any study information that is part of that record. The research team is not required to release research information to you that is not part of your medical record.

Do you need to give the researchers permission to obtain, use or share your PHI? NO! If you decide not to let the research team obtain, use or share your PHI, you should not sign this form, and you will not be allowed to volunteer in the research study. If you do not sign, it will not affect your treatment, payment, or enrollment in any health plans or affect your eligibility for benefits.

# Can you change your mind?

If you decide to stop being in the study, please contact the Lead Researcher or the research staff.

-----FOR IRB USE ONLY------

Rev 11.11.2022 (Amendment 1-03.09.2023)



## 


The research team may ask you whether they can continue to collect information from your medical record. You will also have to decide if you wish to limit the continued use of the information collected during the study. Under US privacy laws you may also withdraw your permission for the researchers to use and share any of your protected information for research, but <u>you must do so in writing</u> to the Lead Researcher at the address on the first page.

Even if you withdraw your permission, the Lead Researcher may still use the information that was already collected, but only to complete this research study. Your health information may still be used or shared after you withdraw your authorization if you have an adverse event (a bad effect) from taking part in the research study.

If you have not already received it, you will also be given The Hospital's Notice of Privacy Practices that contains more information about how The Hospital uses and discloses your PHI.

It is important for you to understand that once information is disclosed to others outside Mount Sinai, the information may be re-disclosed and will no longer be covered by the federal privacy protection regulations. However, where possible, Mount Sinai has entered into agreements with those who will receive your information to continue to protect your confidentiality.

If researchers are reviewing your medical records or asking questions about your medical history or conditions, it is possible that they may learn information related to your HIV status. If that is the case, the following information concerns you. If researchers are not reviewing your medical records or asking questions about your medical history or conditions, then you may ignore the following section.

#### **Notice Concerning HIV-Related Information**

If you are authorizing the release of HIV-related information, you should be aware that the recipient(s) is (are) prohibited from re-disclosing any HIV-related information without your authorization unless permitted to do so under federal or state law. You also have a right to request a list of people who may receive or use your HIV-related information without authorization. If you experience discrimination because of the release or disclosure of HIV-related information, you may contact the New York State Division of Human Rights at (888) 392-3644 or the New York City Commission on Human Rights at (212) 416-0197. These agencies are responsible for protecting your rights.

### How the Institutional Review Board (IRB) can help you:

This research has been reviewed and approved by an Institutional Review Board (IRB). You may reach a representative of the Mount Sinai Program for Protection of Human Subjects at telephone number (212) 824-8200 during regular work hours (Monday-Friday, 9am-5pm, excluding holidays) for any of the reasons listed below. This office will direct your call to the right person within the Mount Sinai Health System:

------FOR IRB USE ONLY------

Rev 11.11.2022 (Amendment 1-03.09,2023)



# 


- Your questions, concerns, or complaints are not being answered by the research team.
- You cannot reach the research team.
- You are not comfortable talking to the research team.
- You have questions about your rights as a research participant.
- You want to get information or provide input about this research.

| FOR IRB USE ONLY |
|------------------|





# 


| Signature of Participant | Printed Name of Participant | Date | Time |
|---|---|---|---|
| PERSON EXPLAINING STUDY | AND OBTAINING CONSENT: | | |
| Signature of Consent Delegate | Printed Name of Consent Delegate | Date | Time |
| WITNESS SECTION: | | | |
| information was accurately expla | hat the information in the consent docun<br>ained to, and apparently understood by, t | | |
| information was accurately explaced consent was freely given by the | ained to, and apparently understood by, t | | |
| consent was freely given by the | ained to, and apparently understood by, t | | |
| consent was freely given by the | ained to, and apparently understood by, t<br>participant. | he participa | ant, and that |
| | ained to, and apparently understood by, t<br>participant. | he participa | ant, and that |

